CLINICAL TRIAL: NCT06786962
Title: Effects of a Virtual Reality Hypnosis Intervention on Reducing Stress and Compassion Fatigue in Neonatal Intensive Care Nurses
Brief Title: Virtual Reality Hypnosis and Nurses' Stress
Acronym: HYPNOVRNEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CARESP: Cellule d'animation régionale en soins palliatifs (Other)
Collaborators: University of Rennes 2 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HYPNOVR - NEONAT
Record Dates: First submitted 2024-12-16; First posted 2025-01-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Hypnosis; Virtual Reality Therapy; Stress; Compassion Fatigue; Compassion Satisfaction; Emotions; Anxiety
Keywords: Hypnosis; Virtual reality; Stress; Compassion fatigue; Neonatal intensive care nurses; Stress reduction program; Non Pharmacological Intervention
MeSH Terms: conditions — Compassion Fatigue; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Neonatal Intensive Care Unit (NICU) Nurses (n = 42) will be randomly assigned to one of two conditions (control or Virtual Reality Hypnosis (VRH)). Each nurse will receive six 10-minute sessions of one of the techniques for 6 weeks (1 session per week).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Participants are seated in a quiet area of the unit. The control group of 21 participants consists of a break with the following instructions and suggestions:
  "Take advantage of this break, this time just for you, to recharge your batteries. Sit in this armchair and I suggest you think of something pleasant and comfortable".
  Interventions: Other: Control arm (SEQ):
- VRH Group (Experimental): The experimental group of 22 participants consists of a hypnosis intervention using a virtual reality device (HypnoVR®).
  Participants are seated in a quiet area of the unit:
  They choose a visual scenario from among 3 proposals, guaranteeing the conditions of a restorative environment. During each session, the same script (support mode) is spoken and the same music (serenity program with soothing tones) is associated with the script. Each participant is fitted with a virtual reality mask and a headset with active noise reduction.
  Interventions: Device: Virtual reality Hypnosis

INTERVENTIONS:
Device: Virtual reality Hypnosis — The experimental group of 22 participants consists of a hypnosis intervention using a virtual reality device (HypnoVR®).
  Participants are seated in a quiet area of the unit:
  They choose a visual scenario from among 3 proposals, guaranteeing the conditions of a restorative environment. During each session, the same script (support mode) is spoken and the same music (serenity program with soothing tones) is associated with the script. Each participant is fitted with a virtual reality mask and a headset with active noise reduction.
  Arms: VRH Group
Other: Control arm (SEQ): — Restoration time
  Participants are seated in a quiet area of the unit. The control group of 21 participants consists of a break with the following instructions and suggestions:
  "Take advantage of this break, this time just for you, to recharge your batteries. Sit in this armchair and I suggest you think of something pleasant and comfortable".
  Arms: Control group

SUMMARY:
The practice of nursing is based on helping relationships and empathy. The work is physically, mentally and emotionally demanding. This requires the mobilization of personal resources (lifestyle, coping strategies) and work resources (managerial, medical support, recognition) to cope with stress. When these resources are present, nurses can activate a resilience process through coping strategies. However, stress levels and emotional impact are such that they can lead to states of suffering and trauma such as compassion fatigue (CF). The prevalence of CF is high in the nursing profession and particularly among neonatal intensive care (NICU) nurses.

Several levels of intervention exist to prevent CF in services: organizational, inter-individual and individual. At the individual level, certain interventions such as meditation have been studied, showing positive effects with the highest levels of evidence.

On the other hand, interventions such as hypnosis have not yet been studied in this context. There is, however, an interest in studying hypnosis as a non-pharmacological intervention to reduce stress and improve emotional regulation. Indeed, the hypnotic process (promoting attentional and cognitive rest, redirecting attentional focus, reducing mental effort) is a resource activator. In order to combine individual and organizational support, the intervention must be offered in the workplace and during working hours, given the difficulty nurses have in extracting themselves from the service, the restricted break time and the acceptability of the virtual reality system. In a context where break time is short and precious, it is necessary to use a tool that adapts to these constraints. Virtual reality with the HypnoVR® tool meets these needs. This device acts as a restorative environment. It has already proven its effectiveness in the care of painful and stressed patients in critical situations. It has not yet been studied in the context of work-related stress in healthcare professionals, such as neonatal intensive care nurses. The protocol takes into account the results of studies reporting the effects associated with the use of virtual reality (VR).

ELIGIBILITY:
Inclusion Criteria:

* Nurse
* Regularly work in a neonatal intensive care unit
* Be of legal age and not opposed to participating in research
* Fluency in French

Exclusion Criteria:

* Age < 18
* Refusal to participate
* Current anticonvulsant or psychotropic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Stress levels | From enrollment to the end of treatment at 8 weeks
  Perceived stress: a single question on stress symptoms : "Stress is a situation in which a person feels tense, restless, nervous or anxious, or can't sleep at night because their mind is constantly troubled. Are you feeling this type of stress these days?" The answer will be recorded on a five-point Likert scale ranging from 1 (not at all) to 5 (a lot).
Emotions | From enrollment to the end of treatment at 8 weeks
  Emotions : 10 items from the short version of the Positive and Negative Affects Schedule .
Anxiety | From enrollment to the end of treatment at 8 weeks
  State anxiety : 10 items from the short version of the State Anxiety Scale
Restoration | From enrollment to the end of treatment at 8 weeks
  Restoration: 3 items from the Mental Restoration Scale
Satisfaction and compassion fatigue | From enrollment to the end of treatment at 8 weeks
  Satisfaction and compassion fatigue: 21 items from the ProQOL - 21 scale
Comfort level | From enrollment to the end of treatment at 8 weeks
  Comfort: indicator of parasympathetic changes in emotional situations during each session, with the ANI Guardian® device.

SECONDARY OUTCOMES:
Evaluation of experience | From enrollment to the end of treatment at 8 weeks
  Experience Open-ended question about the user experience during the session ("Your comments on the session"): "How did you experience this session?" Responses will be analyzed using an approach combining inductive coding and content analysis based on hypnosis processes identified in the literature
Acceptability | From enrollment to the end of treatment at 8 weeks
  To assess acceptability, participants will rate their perception of the relaxation activity using five items from the Unified Theory of Acceptance and Use of Technology (UTAUT). These items assess ease of use, usefulness, effectiveness, overall satisfaction and behavioral intention. Participants will respond on a 10-point Likert scale ranging from 1 (strongly disagree) to 10 (strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Estelle MICHINOV, PhD, Study Director — University of Rennes 2
Locations (1):
- RENNES, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nukarinen, T., Istance, H. O., Rantala, J., Mäkelä, J., Korpela, K., Ronkainen, K., Surakka, V., & Raisamo, R. (2020). Physiological and Psychological Restoration in Matched Real and Virtual Natural Environments. Extended Abstracts of the 2020 CHI Conference on Human Factors in Computing Systems, 1-8. https://doi.org/10.1145/3334480.3382956
- [Result] Asadollah F, Nikfarid L, Sabery M, Varzeshnejad M, Hashemi F. The Impact of Loving-Kindness Meditation on Compassion Fatigue of Nurses Working in the Neonatal Intensive Care Unit: A Randomized Clinical Trial Study. Holist Nurs Pract. 2023 Jul-Aug 01;37(4):215-222. doi: 10.1097/HNP.0000000000000590. PMID 37335149
- [Result] Boselli, E. (2018). Intérêt du monitorage du tonus parasympathique relatif par Analgesia/Nociception Index (ANI) chez les patients anesthésiés ou conscients. Douleurs : Évaluation - Diagnostic - Traitement, 19(5), 205-210. https://doi.org/10.1016/j.douler.2018.07.008
- [Result] Bresesti I, Folgori L, De Bartolo P. Interventions to reduce occupational stress and burn out within neonatal intensive care units: a systematic review. Occup Environ Med. 2020 Aug;77(8):515-519. doi: 10.1136/oemed-2019-106256. Epub 2020 Mar 4. PMID 32132183
- [Result] Figley, C. R. (Éd.). (2015). Compassion fatigue : Coping with secondary traumatic stress disorder in those who treat the traumatized. Routledge.
- [Result] Jess G, Pogatzki-Zahn EM, Zahn PK, Meyer-Friessem CH. Monitoring heart rate variability to assess experimentally induced pain using the analgesia nociception index: A randomised volunteer study. Eur J Anaesthesiol. 2016 Feb;33(2):118-25. doi: 10.1097/EJA.0000000000000304. PMID 26266775
- [Result] Kaplan, S. (1995). The restorative benefits of nature : Toward an integrative framework. Journal of environmental psychology, 15(3), 169-182.
- [Result] Joinson C. Coping with compassion fatigue. Nursing. 1992 Apr;22(4):116, 118-9, 120. No abstract available. PMID 1570090
- [Result] Liang, L., Gobeawan, L., Lau, S.-K., Lin, E. S., & Ang, K. K. (2024). Urban Green Spaces and Mental Well-Being : A Systematic Review of Studies Comparing Virtual Reality versus Real Nature. Future Internet, 16(6), Article 6. https://doi.org/10.3390/fi16060182
- [Result] Ruysschaert, N. (2009). (Self) hypnosis in the prevention of burnout and compassion fatigue for caregivers : Theory and induction. Contemporary Hypnosis (John Wiley & Sons, Inc.), 26(3), 159-172. https://doi.org/10.1002/ch.382
- [Result] Touloudi E, Hassandra M, Galanis E, Goudas M, Theodorakis Y. Applicability of an Immersive Virtual Reality Exercise Training System for Office Workers during Working Hours. Sports (Basel). 2022 Jun 29;10(7):104. doi: 10.3390/sports10070104. PMID 35878115
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Wong JQH, Charles JS, Mok HT, Tan TSZ, Amin Z, Ng YPM. Experiences of healthcare personnel with death in the neonatal intensive care unit: a systematic review of qualitative studies. Arch Dis Child Fetal Neonatal Ed. 2023 Nov;108(6):617-622. doi: 10.1136/archdischild-2023-325566. Epub 2023 May 17. PMID 37197908
- [Result] Zhang YY, Zhang C, Han XR, Li W, Wang YL. Determinants of compassion satisfaction, compassion fatigue and burn out in nursing: A correlative meta-analysis. Medicine (Baltimore). 2018 Jun;97(26):e11086. doi: 10.1097/MD.0000000000011086. PMID 29952947
- [Result] Singer T, Klimecki OM. Empathy and compassion. Curr Biol. 2014 Sep 22;24(18):R875-R878. doi: 10.1016/j.cub.2014.06.054. PMID 25247366
- [Result] Ruiz-Fernandez MD, Perez-Garcia E, Ortega-Galan AM. Quality of Life in Nursing Professionals: Burnout, Fatigue, and Compassion Satisfaction. Int J Environ Res Public Health. 2020 Feb 15;17(4):1253. doi: 10.3390/ijerph17041253. PMID 32075252
- [Result] Boselli E, Musellec H, Bernard F, Guillou N, Hugot P, Augris-Mathieu C, Diot-Junique N, Bouvet L, Allaouchiche B. EFFECTS OF CONVERSATIONAL HYPNOSIS ON RELATIVE PARASYMPATHETIC TONE AND PATIENT COMFORT DURING AXILLARY BRACHIAL PLEXUS BLOCKS FOR AMBULATORY UPPER LIMB SURGERY:A Quasiexperimental Pilot Study. Int J Clin Exp Hypn. 2018 Apr-Jun;66(2):134-146. doi: 10.1080/00207144.2018.1421355. PMID 29601275
- See also: Related Info — https://doi.org/10.1016/j.douler.2018.07.008